CLINICAL TRIAL: NCT00402662
Title: A Phase II Study of Everolimus in Combination With Imatinib in Metastatic Melanoma
Brief Title: A Study of Everolimus in Combination With Imatinib in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unexpected level of toxicity
Sponsor: Yale University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0508000541
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Melanoma
Keywords: everolimus; imatinib
MeSH Terms: conditions — Melanoma | interventions — Everolimus; Imatinib Mesylate

INTERVENTIONS:
Drug: everolimus
Drug: Imatinib

SUMMARY:
The purpose of this study is to determine if the combination of everolimus and imatinib will slow the growth of or cause a reduction in the size of the cancer, and to determine the side effects of the combination in patients with melanoma. Each of the drugs in this combination, if used alone, would not be expected to have an effect against the cancer. However, when used together, there is a possibility that they could work together to damage the cancer cells, or to block the formation or function of the blood vessels that feed the cancer, either of which could result in slowing the growth of or shrinking the cancer. Both drugs work by blocking signals that are sent from outside of a cell to the inside of the cell that direct the cell to make certain substances to keep the cell alive. Cancer cells or blood vessels that feed cancer cells may be more sensitive to drugs that block these signals.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed stage III unresectable or stage IV metastatic melanoma. Patients must have measurable disease as defined by RECIST criteria.
* Patients with up to 1 prior cytotoxic regimen for metastatic disease will be eligible. There will be no prior limitation on adjuvant therapies for stage II/III disease or for patients with stage IV disease treated after resection of all metastatic disease. There will be no prior limitation on biological or hormonal therapies (immune therapies, interferon, hypomethylating agents, histone deacetylase inhibitors, etc.), however, patients previously treated with mTOR inhibitors will be excluded. Prior treatment for metastatic disease is not required. Patients must have recovered from the acute toxicities of prior treatment. Chronic toxicities must have recovered to ≤ grade 1. The minimum interval between prior treatment and first day of dosing on this trial is as follows: standard cytotoxic agents and radiation therapy, 21 days; mitomycin and nitrosoureas, 6 weeks; hormonal and immunotherapy agents, 2 weeks; minor surgery, 2 weeks, major surgery, 3 weeks; investigational agents 4-weeks.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of everolimus in combination with imatinib in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric phase 1 combination trials.
* ECOG performance status < 1.
* Life expectancy of greater than 3 months.
* Patients must have organ and marrow function as defined below:
* Leukocytes >3,000/μL; Absolute neutrophil count >1,500/ μL; platelets >100,000/ μL; Hemoglobin ≥ 9.0 gm/dL (may be transfused to this level); PT/PTT < 1.5x upper limit of normal; Total bilirubin ≤ 2.0 mg/dL;AST(SGOT)/ALT(SGPT) <3X institutional upper limit of normal; Creatinine ≤ 2.0 mg/dL or creatinine clearance >50 mL/min/1.73m2
* The effects of everolimus and imatinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 3 months after stopping study drug. Should a woman (or the partner of a man participating in this trial) become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents. Patients may not have received prior treatment for their cancer with an mTOR inhibitor.
* Patients with known brain metastases or leptomeningeal disease are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with previously treated brain metastases, who no longer require steroids, and have no evidence of progression for at least 8 weeks following treatment of known brain metastases, are eligible.
* Baseline diastolic blood pressure > 95 mmHg. Blood pressure medications may be used to bring the diastolic pressure to levels acceptable for protocol enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular cardiac arrhythmia, myocardial infarction within the previous 6 months, dyspnea at rest, active GI bleeding or ulcer disease, diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because everolimus and imatinib are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with everolimus and imatinib, breastfeeding should be discontinued if the mother is treated on this protocol. These potential risks may also apply to other agents used in this study.
* Known HIV-positive patients, because of the potential for pharmacokinetic interactions with everolimus and imatinib, and because the potential immunosuppressive actions of everolimus may increase progression or infectious complications of HIV. Appropriate studies will be undertaken in HIV-positive patients when indicated.
* Patients receiving warfarin (see section 5.2), or chronic treatment with steroids or another immunosuppressive agent. In addition, patients requiring the following agents are excluded from the study, and must not take the agents while on the trial: ketoconazole, itraconazole, erythromycin, clarithromycin, dexamethasone, phenytoin, carbamazepine, rifampin, Phenobarbital, St. John's Wort, simvastatin, other HMG-CoA reductase inhibitors (if metabolized by CYP3A4), cyclosporine, pimozide, triazolo-benzodiazepines, dihydropyridine calcium channel blockers, and acetaminophen or acetaminophen containing products such as Percoset or Vicodin. Patients taking CYP3A4 interacting agents with narrow therapeutic windows will be excluded from the trial.
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not a allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rate (as defined by RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States